CLINICAL TRIAL: NCT04383496
Title: I CARE for Vets: InCreasing Activity & REcovery for Veterans With PTSD
Brief Title: Increasing Activity for Veterans With PTSD
Acronym: I CARE for Vet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3302-P; RX003302-01A1 (Other Grant/Funding Number: VA RR&D)
Record Dates: First submitted 2020-04-29; First posted 2020-05-12 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD; Exercise; Physical Performance; Mobility Limitation; Wearable Electronic Devices
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Motor Activity; Mobility Limitation | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The intervention uses Graded Exercise Therapy to increase perceived behavioral control by enhancing knowledge about appropriate activities and helping participants set appropriate and attainable daily goals for physical activity. We will also incorporate motivational interviewing techniques and mHealth to enhance positive personal attitudes about physical activity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physical Activity (Experimental): In-person, virtual conferencing, and telephone sessions, wearable device for daily feedback and motivation
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — In-person, virtual conferencing, and telephone sessions, wearable device for daily feedback and motivation

SUMMARY:
The proposed work will be a key step forward in fulfilling the mission of VA RR&D to restore function and enable social reintegration for Veterans. Development of an intervention to increase physical activity may improve physical functioning for Veterans with posttraumatic stress disorder (PTSD), thus addressing an important gap in existing care. If demonstrated to be efficacious in a future randomized trial, this intervention could be implemented throughout VHA to improve quality of life and enable a full recovery for many Veterans with PTSD. Results from the proposed work may also advance our understanding of how to optimally incorporate mobile health technology (mHealth) with more traditional types of patient contacts, such as in-person visits and telephone calls. Effective use of mHealth may offer greater flexibility for VHA clinics looking to implement new programs. Incorporation of mHealth may also increase access to clinical services for Veterans who reside far from VHA facilities.

DETAILED DESCRIPTION:
Veterans with posttraumatic stress disorder (PTSD) have poor physical functioning and there are no existing interventions that effectively address this problem. Our long-term goal is to develop and implement effective interventions to improve physical functioning and reduce risk for adverse health outcomes for Veterans with PTSD. The overall objectives of the proposed project are to develop and pilot test a novel intervention aimed at initiating and maintaining higher levels of physical activity for Veterans with PTSD. This new intervention will address attitudinal and behavioral barriers to increasing physical activity for Veterans with PTSD. Particularly relevant barriers for those with PTSD may include low perceived behavioral control for making positive long-term lifestyle changes and personal attitudes about the harms (vs. benefits) of physical activity.

The proposed work will meet two specific aims: 1) Adapt graded exercise therapy (GET) and incorporate motivational interviewing and mobile health technology (mHealth) to increase physical activity for Veterans with PTSD; and 2) conduct a pilot study to examine the feasibility and acceptability of the intervention for a future randomized controlled trial. To achieve Aim 1, we will develop treatment manuals, training procedures for interventionists, and processes for assessment of intervention fidelity. The intervention will use GET to increase perceived behavioral control by enhancing knowledge about appropriate activities and helping participants set appropriate and attainable daily goals for physical activity. We will also incorporate motivational interviewing techniques and mHealth to enhance positive personal attitudes about physical activity. We will work with our Veteran Engagement Panel for PTSD to refine topics and communication materials. In Aim 2, we will enroll 3 groups of 6-8 participants (18-24 total) and use a concurrent mixed-methods approach to rapidly assess feasibility and acceptability. Quantitative measures will include recruitment (proportion enrolled out of total eligible); attendance (proportion who attend 75% of in-person visits); and retention (proportion who complete post-intervention data collection). Qualitative assessment will consist of semi-structured interviews on acceptability of intervention components (eg, format and topics of in-person visits, usability of mHealth), and barriers and facilitators to attendance. At baseline, during, and post-intervention, we will also measure overall and physical functioning, and collect data on other clinical variables (PTSD symptoms, depressive symptoms, pain, fatigue, and sleep quality) to inform a future effectiveness trial.

The proposed work is innovative because it is a novel combination of GET, motivational interviewing, and mHealth to increase physical activity. It will also be the first intervention to focus on changing physical activity as a means to improving physical functioning for individuals with PTSD. Successful experiences with this program may also help participants build confidence about their general ability to make positive changes related to health, thus increasing the likelihood they will engage in (and adhere to) mental health treatments. If such synergy is ultimately demonstrated, it will open a new direction for VA RR&D and VHA clinical care by indicating that interventions focusing on physical functioning should be more closely integrated with mental health services. Additionally, this project will be one of the first to collaborate with our Veteran Engagement Panel on PTSD research. The format of our panel is adapted from and builds upon previous models of patient stakeholder engagement. Our model addresses many of the barriers to effective stakeholder engagement, including challenges to timely recruitment of patients with relevant experiences, and lack of facilitation expertise among investigators. Completion of this project will help establish the utility of our model of Veteran stakeholder engagement for rapidly developing effective interventions with improved feasibility and acceptability. Thus, this work will enable incorporation of Veteran engagement in future VA research projects.

ELIGIBILITY:
Inclusion Criteria:

* 3 on Primary Care PTSD Screen (PC-PTSD-5)
* "yes" to 3 questions about health-related functional limitations from the Veterans RAND 36-Item Health Survey
* has device and internet access for participating in meetings by videoconference

Exclusion Criteria:

* active suicidal ideation or psychosis
* medical contraindication to participation (eg, complete paraplegia)
* self-reported impairments in 2 or more activities of daily living
* will be permanently moving out of area in next 4 months
* schizophrenia
* acute mental health crisis within the past 3 months (requiring an ED visit or hospitalization)
* routinely completing 150 minutes or more of moderate to vigorous activity per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Denise Duan-Porter, MD PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Goal recruitment was 6-8 participants for each of 3 pilot groups (max 24 total). The actual number of participants enrolled reflects those who completed informed consent and attended the baseline assessment and education session with the physical therapist (6, 8, and 7 for 3 groups). Because this was a group intervention, if participants failed to attend the informed consent or baseline visit (including attempts at rescheduling), we were unable to recruit additional participants for that group.
Pre-assignment Details: 24 participants completed informed consent and were enrolled but only 21 completed the baseline visits (required before moving onto the intervention)
Period: Overall Study
Arm/Group | Physical Activity
Started | 21
Completed | 19
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Physical Activity
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 13
  Race/Ethnicity: Black | 5
  Race/Ethnicity: Asian or Native Hawaiian | 2
  Race/Ethnicity: Hispanic/Latino | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Recruitment
Description: total participants enrolled in intervention (out of total patients identified as eligible)
Time Frame: 2 months
Population: Data represents the total number of participants who completed informed consent
Measure: Count of Participants; unit: Participants
Arm/Group | Physical Activity
Number analyzed (Participants) | 212
Participants | 24

2. Secondary Outcome: Total # Participants Completing Acceptability Interviews
Description: Number of participants who completed interviews on usability of wearable device; barriers and facilitators to attendance
Time Frame: 4 months
Population: Participants who enrolled in study and were invited to interviews
Measure: Count of Participants; unit: Participants
Arm/Group | Physical Activity
Number analyzed (Participants) | 21
Participants | 19

3. Secondary Outcome: Attendance
Description: Number of participants who attended 75% of session visits (3 out of 4 group sessions; 5 of 7 individual follow-up calls)
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Physical Activity
Number analyzed (Participants) | 21
Participants
  Attendance at Group Sessions | 19
  Attendance at Individual Follow-up | 20

4. Secondary Outcome: Retention
Description: Number of participants who complete post-intervention assessments at 4 months follow-up
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Physical Activity
Number analyzed (Participants) | 21
Participants | 17

5. Other Pre Specified Outcome: Physical Activity
Description: Activity tracking (wearable device), number of days meeting activity goal (per week) at 8 weeks
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: days meeting activity goal/week
Groups:
- Intervention Group: Participants who received intervention
Arm/Group | Intervention Group
Number analyzed (Participants) | 19
days meeting activity goal/week | 3.41 (1.85)

6. Other Pre Specified Outcome: Physical Functioning
Description: Physical Component Score of Veterans Short-Form 36 item survey; range 0-100 (standardized), higher is better functioning
Time Frame: 4 months
Population: Participants who completed 4 months follow-up surveys
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 9
units on a scale | 30.9 (5.7)

7. Other Pre Specified Outcome: PTSD Symptoms
Description: PTSD Checklist for DSM V; range 0-80, higher is more symptoms (worse)
Time Frame: 4 months
Population: Complete baseline and follow-up data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Physical Activity
Number analyzed (Participants) | 17
units on a scale | 49.6 (16.1)

8. Other Pre Specified Outcome: Depressive Symptoms
Description: Patient health questionnaire 8-item; range 0-24, higher is more symptoms (worse)
Time Frame: 4 months
Population: complete follow-up data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Physical Activity
Number analyzed (Participants) | 16
units on a scale | 7.63 (5.54)

9. Other Pre Specified Outcome: Pain Intensity and Interference
Description: PEG (brief 3-item scale on intensity and interference), range 0-10, higher is more pain/interference
Time Frame: 4 months
Population: complete follow-up data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Physical Activity
Number analyzed (Participants) | 16
units on a scale | 5.1 (2.1)

10. Other Pre Specified Outcome: Fatigue
Description: Patient Reported Outcomes Measurement Information System (PROMIS) fatigue 4-item short form, range 0-100 (standardized), higher is more fatigue
Time Frame: 4 months
Population: participants with complete follow-up data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Activity
Number analyzed (Participants) | 15
score on a scale | 55.8 (11.2)

11. Other Pre Specified Outcome: Sleep-related Impairment
Description: PROMIS sleep measure, standardized T score (0-100), higher is poorer sleep
Time Frame: 4 months
Population: complete follow-up data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Activity
Number analyzed (Participants) | 15
score on a scale | 56.7 (11.2)

12. Other Pre Specified Outcome: 6 Minute Walk
Description: distance walked in 6 min (in meters)
Time Frame: 4 months
Population: complete follow-up data
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Physical Activity
Number analyzed (Participants) | 17
meters | 539 (114)

13. Other Pre Specified Outcome: Sit to Stand
Description: # of sit-to-stands completed in 30 seconds
Time Frame: 4 months
Population: complete follow-up data
Measure: Mean (Standard Deviation); unit: sit-to-stand events
Arm/Group | Physical Activity
Number analyzed (Participants) | 17
sit-to-stand events | 19.1 (9.6)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Physical Activity
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Activity (N=21)
Skin irritation at wrist due to wearing fitness device (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT04383496/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT04383496/ICF_000.pdf